CLINICAL TRIAL: NCT05684315
Title: Effect of Tissue Flossing on Recovery Time After Intense Physical Exercise Causing Delayed Onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Academy of Physical Education
Record Dates: First submitted 2023-01-03; First posted 2023-01-13 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-02

CONDITIONS: Health Behavior; Muscle Strain, Lower Leg
Keywords: health behavior; hamstring flexibility; fascial shearing; delayed onset muscle soreness; muscle disorder; treatment; blood flow restriction training; myotonometer; muscle stiffness
MeSH Terms: conditions — Health Behavior; Sprains and Strains; Muscular Diseases | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two rounds over 4 weeks. In the first round, subjects will have one leg threaded during the fatigue protocol, and after a four-week rest after full recovery, they will have the other leg threaded during the fatigue protocol.
Who Masked: Participant, Investigator
Masking Description: The subjects will not be informed what activity awaits them and which leg will be subjected to intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- soft tissue flossing therapy right lower limb (Experimental): The study will be conducted in two rounds, 4 weeks apart. In round one, subjects will have their right leg flossed while performing the fatigue protocol.
  Interventions: Procedure: soft tissue flossing therapy
- soft tissue flossing therapy left lower limb (Experimental): The study will be conducted in two rounds, 4 weeks apart. In round one, subjects will have their left leg flossed while performing the fatigue protocol.
  Interventions: Procedure: soft tissue flossing therapy

INTERVENTIONS:
Procedure: soft tissue flossing therapy — BFRT and tissue threading is a therapy that involves applying external pressure below or above a joint or muscle of a selected limb, usually with a circumferential elastic band. The pressure provided by the rolled band securely maintains arterial blood supply but reduces or blocks venous outflow distal to the site.
  Other Names: Blood Flow Restriction Training; BFRT

SUMMARY:
The aim of the study is to assess whether soft tissue flossing therapy will alleviate eccentric muscle-destroying influences. Men aged 20-25 will be tested. Suddenly taking up activity in untrained people and performing the fatigue protocol is a heavy burden for the body, and its effects may have a negative impact on the body. The assessment of the processes taking place in the body under the influence of this type of physical activity with the use of soft tissue flossing will broaden the scope of knowledge about this therapeutic method and will allow assessing whether it has an impact on accelerating regeneration after intense physical exertion.

ELIGIBILITY:
Inclusion Criteria:

* men aged 20-25
* BMI (body mass index) at the level of 20-35

Exclusion Criteria:

• chronic diseases, musculoskeletal injuries, mental disorders, surgery or hospitalization

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Isokinetic muscle strength | 40 days
  Measurements will be performed on an isokinetic dynamometer (Biodex Medical System 4-PRO, New York, USA). According to the manufacturer's protocol, the dynamometer will be calibrated before each test session. The gravity correction will be performed before each series of measurements. Before the intervention, participants will perform a 5-minute warm-up on the bicycle ergometer with a power of 120 W.

SECONDARY OUTCOMES:
Soft tissue assessment | 40 days
  Changes in quadriceps femoris stiffness will be assessed by myometry performed separately for six points marked on the muscle before the test.
Range of motion | 40 days
  Knee Range of motion will be measured with a 360° 14- inch hand held metal goniometer (Fabrication Enterprises, USA). During the measurement, the tested person will be in the supine position. A stabilizing belt will be placed at the height of the sacrum. The axis of rotation of the goniometer will be set at the height of the space of the knee joint. One arm of the goniometer will be aimed at the greater trochanter and the other arm at the lateral malleolus of the fibula. Landmarks for subsequent measurements will be marked on the first day on the subjects' bodies with a semi-permanent marker. Participants will be asked to perform maximum full knee flexion. The knee angle measurement will be repeated three times, and the average result will be included in further analysis.
Visual Analogue Scale (1-100 mm) | 40 days
  A Visual Analogue Scale will be was used to assess pain - the subjects will mark the level of pain perception on a colour scale (1-100 mm) immediately after all exercise tests where a value of 1 is attributed to no pain at all, and a value of 100 is the worst pain imaginable.
Pain assessment - Algometer | 40 days
  Measurement of the pain threshold under the influence of pressure on the muscle will be tested with a digital algometer "Digital Force Algometer" at six points marked on the muscle before the tests.
Triple hop jump test | 40 days
  In the triple jump test, subjects will perform the longest possible jump on one leg three times in a row. During the test, they must not lose their balance and must land safely. The distance will be measured from the starting line to the supporting heel.

CONTACTS AND LOCATIONS:
Overall Officials: Szczepan Wiecha, Phd, Study Director — Jozef Pilsudski University of Physical Education in Warsaw Faculty in Biala Podlaska
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw Faculty in Biala Podlaska, Biała Podlaska, Poland